CLINICAL TRIAL: NCT02553122
Title: The Combined Efficacy of Evicel and Tranexamic Acid on Total Knee Arthroplasty During the Early Perioperative Period
Brief Title: The Combined Efficacy of Evicel and Tranexamic Acid on Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Data has been published on this study (this would have been a duplicate study)
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Sun Jin Kim, Chief of Adult Reconstruction, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-12-178
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Blood Loss; Tranexamic Acid; Evicel
MeSH Terms: conditions — Hemorrhage | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Other): This group of patients will receive standard protocol to control intra-operative blood loss.
  Interventions: Device: tourniquet
- Treatment Group (Active Comparator): This group of patients will receive TXA, Evicel and standard protocol to control intra-operative blood loss.
  Interventions: Drug: Evicel

INTERVENTIONS:
Drug: Evicel — Fibrant Sealant to apply on the soft tissue to control intra-operative blood loss
  Arms: Treatment Group
Device: tourniquet — A tourniquet is applied to the thigh to stop/ decrease blood flow
  Arms: Control Group

SUMMARY:
Total knee arthroplasty is a surgical procedure that involves a significant amount of blood loss and it has always been the surgeons' goal to try to minimize blood loss. In the current study, we will investigate the effect of blood loss after total knee arthroplasty with the combination of Evicel, a fibrin sealant and Tranexamic Acid.

DETAILED DESCRIPTION:
Introduction and Background: Total knee arthroplasty is characterized by a large amount of postoperative blood loss and frequent need for blood transfusions.1 Also of concern is the risk of hematomas which can potentially lead to infection or wound complications and delay the overall rehabilitation process.2 By reducing postoperative bleeding, the outcomes of total knee arthroplasty would be improved by better range of motion, less frequency of blood transfusion and decreased incidence of arthrofibrosis.3 Several studies have looked at different blood conservation strategies including reinfusion of drains, tourniquets, autologous blood transfusions, topical and intravenous antifibrinolytic alone, topical fibrin sealant alone, and monopolar and bipolar electrocautery. The combined use of a topical fibrin sealant (Evicel®) with an antifibrinolytic (Tranexamic acid) represents another approach to reducing blood loss in patients undergoing total knee arthroplasty. Evicel® is a fibrin sealant consisting of human-derived thrombin and fibrinogen that work in combination to form a stable blood clot at the bleeding site. Evicel® is regularly used in orthopaedic and other sub-specialty surgeries. One investigation has reported on the use of a topical hemostatic agent in total knee arthroplasty.4 It compared the use of a fibrin sealant for hemostasis with standard hemostasis protocols and found that the topical hemostatic agent decreased post operative blood loss, increased post operative hemoglobin levels, and resulted in a decrease in the need for post operative blood transfusion. Tranexamic Acid is given topically or intravenously to occlude the fibrin cleavage sites on plasminogen and inhibit the breakdown of fibrin clots. Tranexamic acid is also regularly used in orthopaedic and other sub-specialty surgeries. Studies have found that intravenous dosing of tranexamic acid prior to incision, and again after tourniquet release reduces the need for the blood transfusion versus standard hemostasis.5, 6

Research Questions/Objectives: Does the combination use of a fibrin sealant and an antifibrinolytic in our institutional total knee arthroplasty protocol decrease postoperative drain output/hematocrit drop/hemoglobin drop or the need for post operative blood transfusions compared to standard hemostasis technique? Secondary objectives will be measuring differences in postoperative pain, postoperative range of motion, and rates of postoperative complications including pulmonary embolism, deep vein thrombosis, and wound complications requiring a return to the operating room between treatment and control groups.

Study Design: The null hypothesis states that the combined use of a topical fibrin sealant and an antifibrinolytic in total knee arthroplasty will show no difference in the amount of postoperative blood loss compared to the standard means of hemostasis (tourniquet and electrocauterization). The study will be a prospective randomized trial with patients that are undergoing elective primary, unilateral, cemented total knee arthroplasty. Patients will be randomly divided into two groups. A control group, in which the standard means of hemostasis will be applied and a treatment group, in which the standard means of hemostasis will be applied with the additional use of Evicel® (a fibrin sealant) and Tranexamic acid (an antifibrinolytic). All operations will be standardized between four surgeons.

Subjects: The target population is patients seen in the outpatient office who are indicated for primary total knee arthroplasty. Patients will be asked if they would like to participate in the study; only patients capable of consenting to surgery will be enrolled. Patients undergoing total knee arthroplasty revisions and patients with blood disorders, on chronic anti-thrombotic medication such as Coumadin and any patients with a history of deep vein thrombosis and/or pulmonary embolism will be excluded. Despite that Evicel® contains human-derived blood products, Jehovah's Witnesses will not be excluded and these patients will be given an opportunity whether they would like to participate or not. As tranexamic acid is renally cleared, renally impaired individuals will be excluded.

Study Procedures: All participating surgeons will adhere to the same protocol. Upon enrolling in the study, patient demographics including age, gender, height, weight will be recorded and stored in an encrypted, protected database. Eligible / consenting patients will be randomized in a 1:1 ratio to receive either treatment or non-treatment. The randomization will be stratified by surgeon to ensure balanced assignment of treatment / non-treatment in each of participating surgeons. Randomization schemes will be generated and maintained by Dr. David Leibelt, the study statistician. Dr. Leibelt will provide Mr. Bharat Tiwari with a set of randomization envelopes to be stored and used in the study clinic. Mr. Tiwari will assign these envelopes in sequential order, by envelope number and surgeon, to eligible /consenting patients. . During the process, Dr. Jason Wong and Mr. Andrew Schwartz will be blinded and will have no access to the randomization assignment. Preoperative blood work including hematocrit and hemoglobin will be performed, a standard for patients undergoing joint arthroplasty. On the day of surgery, the patients will be seen in the preoperative holding area, and again be asked if they consent to take part in the study. Total knee arthroplasty will then be performed with a standard medial parapatellar approach using a 350 mm Hg pneumatic tourniquet on the operative leg. All surgeons will use Zimmer implants. After patient is put to sleep, attending surgeon will inform the operating team that whether the patient is randomized into the treatment or control group. If the patient is part of the treatment group, they will receive a 10 mg/kg dose of tranexamic acid prior to tourniquet inflation. After removal of trial implants and irrigation/thorough drying, 2 mL of Evicel® will be sprayed (under 15-25 psi of CO2) into the posterior joint capsule (via the gap between femur and tibia). Once the implants are in place and the methylmethacrylate cement is cured, the joints will be irrigated copiously and dried thoroughly for the final time. 2 mL of Evicel® will be dripped into pinholes, another 2 mL of Evicel® will be dripped along the exposed edges of bony tissue, and an additional 2 mL of Evicel® will be sprayed on all remaining soft tissue. After 2 minutes, the tourniquet will be released and a second dose of 10 mg/kg tranexamic acid will be given as electrocautery is being performed. After joint capsule closure, a final 2 mL of Evicel® will be sprayed along the arthrotomy incision and on subcutaneous soft tissue. On top of the treatment protocol mentioned above, patient will also receive the standard tourniquet protocol and electrocautery. If the patient is in the control group, the standard tourniquet protocol and electrocautery alone will be used for hemostasis. In both groups, an auto transfusion drain will then be placed within the deep layer of the knee. The joint will then be closed and dressed in standard fashion. The patient will then be taken to the postoperative anesthesia care unit. Immediate postoperative hemoglobin and hematocrit levels will be recorded, a standard practice at our institution. The drain output will be recorded over a 24-hour period. As is standard, hemoglobin and hematocrit levels will be recorded for the three days postoperatively. Any transfusions and/or complications (pulmonary embolism, deep vein thrombosis, and wound complications requiring a return to the operating room) and length of stay will be monitored (according to standard protocol) and recorded. Pain scores utilizing the WOMAC, SF-36, and VAS scales will be recorded during postoperative follow up in the clinic. Range of motion will be compared to preoperative values at two and six weeks postoperatively.

Safety outcomes to be monitored

Potential complications associated with the study such as pulmonary embolism, deep vein thrombosis, and wound complications that require a return to the operating room will be monitored by the surgical team.

Risks and Benefits

Potential benefits include decreased perioperative blood loss, which would sequentially decrease the chance of blood transfusion (lower costs, fewer infections and errors, and less frequent seroconversion) and decreased pain secondary to joint hematoma. This study also aims to eliminate the need for post-operative drain usage (lower cost, fewer infections, fewer drain complications and less time in the operating room).

Evicel consists of human-derived thrombin and fibrinogen. Patients with known allergies to human blood products should not participate in this study. Also, the human-derived blood products carry a risk of transmitting infectious agents such as viruses and theoretically, the Creutzfeldt-Jakob disease (CJD) agent. This risk is theoretically equal to the risk of a blood transfusion; however, there have been NO known incidents of infectious agent being transmitted from the use of Evicel. Evicel is FDA approved and routinely used in orthopaedic surgery.

Tranexamic acid is a pro-coagulant molecule that should not be used in patients with a past medical history of intravascular clotting. Dosing of tranexamic acid should be reduced in a renally impaired patient. The compound also should be avoided in those with known allergies to tranexamic acid. Tranexamic acid is FDA approved and routinely used in a variety of surgeries, including orthopaedics

Data Safety Monitoring Plan

A data safety monitoring board consists of an independent physician, Dr. Tony Wanich, Mr. Bharat Tiwari and Dr.Yungtai Lo. At the 50 and 100 patient mark, the board will decide based on the following criteria and decide on whether or not the study should be continued:

1. whether or not the complications rates (includes deep vein thrombosis, cerebrovascular accidents) between the treatment group and the control group is significantly different
2. whether or not the transfusion rates between the treatment group and control group is significantly different
3. whether or not the drain output between the treatment group and the control group is significant different If any of the above criteria is met, the board will inform the principle investigator and decide on whether or not the study should be terminated early.

Data Management and Analysis:

Measures: The primary outcome measured will be 24-hour drain output that will be measured from the time it is introduced. Secondary measures will be the serum hemoglobin and hematocrit levels measured approximately 2 weeks prior to surgery and each of the first three days after surgery. Transfusions throughout the duration of stay and the length of hospital stay will also be recorded. Scores obtained from 3 pain scales will be recorded: WOMAC (Pre-op and Post-op at 6 months), SF-36 (Pre-op and Post-op at 6 months), and VAS (Pre-op, Post-op day # 1, 2, 3, Post-op visit #1 and 2). Range of motion at two and six weeks postoperatively will be compared to the preoperative range. All measurements will be recorded in an encrypted and protected database.

Statistical Analysis: The primary (drain output) and secondary (hemoglobin/hematocrit) outcomes are continuous variables. Values for the intervention (Evicel®/Tranexamic acid) and the standard of care control groups will be compared with the Mann-Whitney test. Results for individual day measures and the summary measures (total drainage and average hemoglobin/hematocrit) will not be adjusted for multiple comparisons. However, if any statistically significant results from different days of the same measure and the composite measure are not consistent, the possibility of type I error will be emphasized. We will assume the data will not be normally distributed and therefore a non-parametric test, Mann Whitney test, will be performed. We expect our randomization to result in balanced study groups in regards to characteristics like age, sex, race, and BMI. Therefore stratified randomization is unnecessary. However, if the two study arms are not reasonably balanced, additional analyses using linear regression adjusting for any unbalanced variables will be performed. Intention to treat analyses will be performed. Statistical analyses will be completed by Dr. Jason Wong and medical student, Andrew Schwartz. Both Dr. Wong and Mr. Schwartz will be blinded about the randomization.

Sample Size: Based on previous studies looking at similar outcomes and using a conservative estimate for true difference of means of drain output, we need 50 patients per group for 90% power and 150 patients per group for 97% power to detect a difference in 24 hour drain output.

Implementation Plan/Timetable: Patients will be seen in the office and, if indicated for total knee arthroplasty, we will request consent for the study. The attending surgeons will answer any question at that time. A physician assistant who is blinded will collect data daily. An average of 15-20 total knee arthroplasties are done each week. The data collection will likely take 3-6 months. The data collected will be kept on an encrypted and protected database accessible only to the physicians caring for the patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee

Exclusion Criteria:

* bleeding disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 3 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jin Kim, MD, Principal Investigator — Montefiore Medical Center

REFERENCES:
- [Result] Levy O, Martinowitz U, Oran A, Tauber C, Horoszowski H. The use of fibrin tissue adhesive to reduce blood loss and the need for blood transfusion after total knee arthroplasty. A prospective, randomized, multicenter study. J Bone Joint Surg Am. 1999 Nov;81(11):1580-8. doi: 10.2106/00004623-199911000-00010. PMID 10565650
- [Result] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147